

| Partici | pant | Study | / ID: |
|---------|------|-------|-------|

## **CONSENT FORM**

A Proof-of-Concept Study to Assess the Efficacy of Symprove Probiotics in Managing Persistent Gastrointestinal Symptoms in Adult Coeliac Disease Patients in Histological Remission

Name of Researcher: [insert CI name]

Please initial box

| | I confirm that I have read and understood the information sheet ([insert |
|---|---|
| 1 | version & date]) for the above study. I have had the opportunity to consider |
| | the information, ask questions and have had these answered satisfactorily. |
| | I understand that my participation is voluntary and that I am free to withdraw |
| 2 | at any time without giving any reason, without my medical care or legal rights |
| | being affected. |
| | I understand that relevant sections of my medical notes and data collected |
| | during the study, may be looked at by individuals from regulatory authorities |
| 3 | or from the NHS Trust, where it is relevant to my taking part in this research. |
| | I give permission for these individuals to have access to my records to make |
| | sure the research has been managed correctly. |
| | I understand that I will take Symprove (70ml daily) for 3 months and |
| 4 | complete questionnaires about my symptoms and quality of life monthly |
| | during this period. |
| | I understand that taking Symprove may cause mild gastrointestinal |
| 5 | discomfort initially, which typically resolves within a few days, and that this is |
| | a widely available food supplement with a good safety profile. |
| | I agree to provide stool samples as part of my involvement in this study at |
| | baseline (Month 0) and Month 3. I understand that these samples will be |
| 6 | labelled with a study ID and not my name, and sent to a commercial |
| | Laboratory (in Europe) to be analysed for gut bacteria and then destroyed, |
| | and that I will not gain any direct personal or financial benefit from them. |
| 7 | I agree to take part in the above study |
| | OPTIONAL: I agree that data collected for this study can be used for future |
| 8 | research and may be shared anonymously with external researchers based |
| | worldwide, as detailed in the information sheet. |



| Signatures: | | | | |
|---|---|---|---|---|
| Name of Part | ticipant | <br>Date | | Signature |
| | son taking consent | | original) to be kept in me | Signature<br>edical notes. |
| Participant Contact Details: | | | | |
| Name: | | | | |
| Address: | | | | |
| Telephone: | | | | |
| Email: | | | | |
| Preferred method of contact for study updates: | | | | |
| | Email | ☐ Post | | ☐ Telephone |
| Would you like to receive a summary of the study results when available? | | | | |
| | □ Yes | П № | | |